CLINICAL TRIAL: NCT05372705
Title: Reducing Eco-anxiety and Increasing Eco-action in Adolescents Using Selfie Videos: a Randomized Controlled Trial
Brief Title: Reducing Eco-anxiety Using Selfies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000028980_d
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Ecology; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive (Active Comparator): ~58-second selfie video (TikTok) of an adolescent presenting a "can do" / climate action / positive perspective on global warming
  Interventions: Behavioral: Short videos
- Negative (Active Comparator): ~58-second selfie video (TikTok) of an adolescent presenting an "it's already too late" / climate catastrophe / negative perspective on global warming
  Interventions: Behavioral: Short videos
- Neutral (Active Comparator): ~58-second selfie video (TikTok) of an adolescent discussing a topic unrelated to climate change or global warming
  Interventions: Behavioral: Short videos

INTERVENTIONS:
Behavioral: Short videos — Intervention videos will each be of 90-second duration and feature four underage professionals (ages 16) acting as simulated patients. All videos will focus on an empowered presenter with depression sharing their personal story regarding depression and describe how social supports from family, friends, and community, as well as professional help assisted them in overcoming symptoms of their illness. The actors will include a transgender male, a cis-gender male, a transgender female, and a cis-gender female.

SUMMARY:
The purposes of this study are to test among adolescent viewers the utility of selfie (TikTok) short video-based interventions to:

1. Reduce ecological anxiety,
2. Increase ecological agency,
3. Compare two different types of messaging, and
4. Examine the role of viewer's gender and race as independent factors on the outcomes of interest.

DETAILED DESCRIPTION:
Intervention videos will each be TikTok self-recorded videos (of 58-second duration) featuring the same underage professional (ages 16) acting as simulated participant. Video 1 ("Negative") will focus on impending ecological catastrophic outcomes; Video 2 ("Positive") will focus on the actions that youth will be able to take in preventing such outcomes; and Video 3 ("Neutral") will include content unrelated to ecological concerns.

We intend to assign ~1,000 individuals aged 14-18 in a randomized way, in equal proportions, and stratified by sex and race, to view one of the three TikTok videos: Positive, Negative, or Neutral.

Assessments will occur at baseline and post-intervention, and will include:

1. Demographics (baseline only),
2. Primary outcome:

   a. Climate Change Anxiety scale (13 items)
3. Secondary outcome:

   1. Climate Hope scale (11 items)
   2. Behavioral intentions (6 items; adapted from)29,
   3. Hopefulness and agency sliders (2 items), and
   4. Three words

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Living in the US
* Ages 14 - 18

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Climate Change Anxiety Scale (CCAS) | Within 10 minutes
  The CCAS is the sum of 13 items (Clayton and Karazsia; Journal of Environmental Psychology, 2020). Each of the items is a statement on which participants are asked to rate their agreement on a 5-point Likert-type scale: from 1 ("Never") to 5 ("Almost always".)
  The range of the scale is from 13 to 65; higher scores indicate greater eco-axiety.

SECONDARY OUTCOMES:
Change in Climate Change Hope Scale (CCHS) | Within 10 minutes
  The CCHS is the sum of 11 items (Li and Moore; Environ Behav, 2018). Each of the items is a statement on which participants are asked to rate their agreement on a 5-point Likert-type scale: from 1 ("Not at all") to 5 ("A great deal".)
  The range of the scale is from 11 to 55; higher scores indicate greater hope regarding environmental action.
Change in Environmental Action Scale-Behavioral Intentions (EAS-BI) | Within 10 minutes
  We will use the Behavioral Intentions component of the Environmental Action Scale (Alisat and Riemer; J Environ Psychol, 2015.) The BI component is the sum of 6 items. Each of the items is a statement on which participants are asked to rate their agreement on a 5-point Likert-type scale: from 1 ("Not at all") to 5 ("A great deal".)
  The range of the scale is from 6 to 30; higher scores indicate greater environmental action behavioral intentions.
Change in Hopefulness "slider" | Within 10 minutes
  Participants will be asked to rate how hopeful they are about global warming. They will move a continuous slider ranging from 0 ("Not hopeful at all; we are doomed regarding global warming and its consequences") to 100 ("Very hopeful; our actions can revert and prevent global warming and its consequences".)
Change in Agency "slider" | Within 10 minutes
  Participants will be asked to rate how much agency they consider having around global warming. They will move a continuous slider ranging from 0 ("There is nothing that I can do about it") to 100 ("There is a lot that I can do about it".)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale Child Center, New Haven, Connecticut
  - Yale Child Study Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin A, Calhoun A, Paez J, Amsalem D. Destigmatizing perceptions about Black adolescent depression: randomized controlled trial of brief social contact-based video interventions. J Child Psychol Psychiatry. 2022 Nov;63(11):1270-1278. doi: 10.1111/jcpp.13570. Epub 2022 Jan 23. PMID 35066880
- [Background] Amsalem D, Martin A. Reducing depression-related stigma and increasing treatment seeking among adolescents: randomized controlled trial of a brief video intervention. J Child Psychol Psychiatry. 2022 Feb;63(2):210-217. doi: 10.1111/jcpp.13427. Epub 2021 Apr 6. PMID 33821507
- [Background] Amsalem D, Halloran J, Penque B, Celentano J, Martin A. Effect of a Brief Social Contact Video on Transphobia and Depression-Related Stigma Among Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220376. doi: 10.1001/jamanetworkopen.2022.0376. PMID 35212749
- [Background] Benoit L, Thomas I, Martin A. Review: Ecological awareness, anxiety, and actions among youth and their parents - a qualitative study of newspaper narratives. Child Adolesc Ment Health. 2022 Feb;27(1):47-58. doi: 10.1111/camh.12514. Epub 2021 Oct 22. PMID 34687125